CLINICAL TRIAL: NCT04725760
Title: Evaluation of the Efficacy of the BrainPort Vision Pro on the Performance of Daily Activities in the Profoundly Blind French Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wicab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-WIFR-8313
Record Dates: First submitted 2021-01-15; First posted 2021-01-27 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-01

CONDITIONS: Blindness
Keywords: blindness; brainport; brainport vision pro; assistive device; assistive technology; visual impairment
MeSH Terms: conditions — Blindness; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Group Assisgnment (Experimental)
  Interventions: Device: BrainPort Vision Pro

INTERVENTIONS:
Device: BrainPort Vision Pro — Ten hours of training over 3 to 5 days, followed by autonomous use of the device.
  It will be recommended that the subject use the BrainPort® Vision Pro device for at least 5 hours per month for a period of 12 months.

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of the BrainPort® Vision Pro, an electronic oral assistive device, in the performance of daily tasks by French persons who have residual vision limited to light perception or less in both eyes.

ELIGIBILITY:
Inclusion Criteria:

1. 8 years of age or older
2. Diagnosis of profound blindness with residual vision limited to a perception of light or lower in both eyes.
3. Minimum post 12 months diagnosis of blindness
4. Previously completed conventional rehabilitation such as orientation and mobility training with a cane or guide dog.
5. Ability to be read and to understand the documentation and procedures of the study.
6. Ability to provide feedback on the use of the BrainPort Vision Pro device.
7. Ability to use basic computer and/or other technologies.
8. Willing and able to answer all questionnaires, carry out telephone follow-ups, undergo device training and carry out all study procedures, after having passed the orientation phase with the device.
9. Participant or his legal representative willing and able to sign informed consent.

Exclusion Criteria:

1. Ongoing oral disorders determined on the basis of the participant's medical history and/or by an examination of the oral cavity by a dental specialist.
2. History of tongue damage resulting in sensitivity problems or impaired language.
3. Visible open sores, herpes, abrasions, blisters or rashes on the tongue or numbness of the tongue.
4. Piercings on the tongue.
5. Planned or recent oral surgery (in the last 3 months) and/or dental care (excluding oral check-ups or routine scaling).
6. Known neuropathy of the language or sensory system.
7. History of seizures or epilepsy.
8. Pregnant woman, willing to be pregnant or lactating. Women of childbearing age should consent to the use of appropriate contraception to avoid pregnancy during the study period.
9. Implanted medical devices (e.g., pacemaker, deep brain stimulation device, cochlear implant).
10. Any hearing impairment that prevents you from hearing the device's announcements.
11. Cognitive impairment detected on the basis of medical history and/or during a cognitive impairment telephone interview.
12. Expected or ongoing participation in another clinical trial or any research that may interfere with this study.
13. Known allergy to nickel, gold or a stainless-steel component.
14. Any health condition that may interfere with the study's evaluations.
15. A person unable to assemble the device and/or interpret the device's signals or who refuses to continue to participate in the study after passing the initial training phase with the device.
16. Person deemed unfit to participate in the study by the lead investigator for any other previously cited reason.
17. Adults who do not have the ability to provide valid informed consent (under legal protection)

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Function | Baseline
  Ultra Low Vision - Visual Function Questionnaire - 50 (ULV-VFQ-50), Aa validated self-assessment scale to measure functional vision in people with ultra low vision. 50 items on a Likert scale, ranging from 1-4, higher scores indicated more difficult (lower visual ability)
Visual Function | 3 months
  Ultra Low Vision - Visual Function Questionnaire - 50 (ULV-VFQ-50), Aa validated self-assessment scale to measure functional vision in people with ultra low vision 50 items on a Likert scale, ranging from 1-4, higher scores indicated more difficult (lower visual ability)
Visual Function | 6 months
  Ultra Low Vision - Visual Function Questionnaire - 50 (ULV-VFQ-50), Aa validated self-assessment scale to measure functional vision in people with ultra low vision 50 items on a Likert scale, ranging from 1-4, higher scores indicated more difficult (lower visual ability)
Visual Function | 12 months
  Ultra Low Vision - Visual Function Questionnaire - 50 (ULV-VFQ-50), Aa validated self-assessment scale to measure functional vision in people with ultra low vision 50 items on a Likert scale, ranging from 1-4, higher scores indicated more difficult (lower visual ability)

SECONDARY OUTCOMES:
Object recognition | Baseline
  Subjects will be asked to reach and grasp one of four objects requested by the examiner, without touching any other object. A total of 10 tests will be conducted. If the test is not answered after two minutes, the test will be considered incorrect. The number of correctly identified objects will be recorded.
Character identification | Baseline
  High contrast letters and numbers will be presented. Subjects will be required to orally identify each letter or number presented. The total number of correct answers will be recorded. Ten individual letters/numbers will be presented.
Orientation and mobility tasks | Baseline
  This task will measure participants' ability to navigate a room and identify distinct objects and features in their environment, such as windows and doorways.
Object recognition | 3 months
  Subjects will be asked to reach and grasp one of four objects requested by the examiner, without touching any other object. A total of 10 tests will be conducted. If the test is not answered after two minutes, the test will be considered incorrect. The number of correctly identified objects will be recorded.
Character identification | 3 months
  High contrast letters and numbers will be presented. Subjects will be required to orally identify each letter or number presented. The total number of correct answers will be recorded. Ten individual letters/numbers will be presented.
Orientation and mobility tasks | 3 months
  This task will measure participants' ability to navigate a room and identify distinct objects and features in their environment, such as windows and doorways.
Object recognition | 6 months
  Subjects will be asked to reach and grasp one of four objects requested by the examiner, without touching any other object. A total of 10 tests will be conducted. If the test is not answered after two minutes, the test will be considered incorrect. The number of correctly identified objects will be recorded.
Character identification | 6 months
  High contrast letters and numbers will be presented. Subjects will be required to orally identify each letter or number presented. The total number of correct answers will be recorded. Ten individual letters/numbers will be presented.
Orientation and mobility tasks | 6 months
  This task will measure participants' ability to navigate a room and identify distinct objects and features in their environment, such as windows and doorways.
Object recognition | 12 months
  Subjects will be asked to reach and grasp one of four objects requested by the examiner, without touching any other object. A total of 10 tests will be conducted. If the test is not answered after two minutes, the test will be considered incorrect. The number of correctly identified objects will be recorded.
Character identification | 12 months
  High contrast letters and numbers will be presented. Subjects will be required to orally identify each letter or number presented. The total number of correct answers will be recorded. Ten individual letters/numbers will be presented.
Orientation and mobility tasks | 12 months
  This task will measure participants' ability to navigate a room and identify distinct objects and features in their environment, such as windows and doorways.
Impact of Vision Impairment-Very Low Vision Quality of Life Scale | Baseline
  A vision-related quality of life scale for participants with very low vision 28 items on a Likert scale, ranging from 1-3 with higher scores indicating better vision-related quality of life.
Impact of Vision Impairment-Very Low Vision Quality of Life Scale, | 3 months
  A vision-related quality of life scale for participants with very low vision 28 items on a Likert scale, ranging from 1-3 with higher scores indicating better vision-related quality of life.
Impact of Vision Impairment-Very Low Vision Quality of Life Scale, | 6 months
  A vision-related quality of life scale for participants with very low vision 28 items on a Likert scale, ranging from 1-3 with higher scores indicating better vision-related quality of life.
Impact of Vision Impairment-Very Low Vision Quality of Life Scale, | 12 months
  A vision-related quality of life scale for participants with very low vision 28 items on a Likert scale, ranging from 1-3 with higher scores indicating better vision-related quality of life.
Adverse events related to device or study procedures | 12 months
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Grant, Ph.D., Study Director — Wicab, Inc.; Isabelle Audo, Ph.D., Principal Investigator — National Hospital for Ophthalmology of the Fifteen-Vingts
Locations (7):
- France (7):
  - University Hospital La Timone, Marseille
  - CHU de Montpellier, Montpellier
  - University Hospital of Nantes, Nantes
  - Institut Aramav, Nîmes
  - Fondation hospitalière Sainte-Marie, Paris
  - Necker-Enfants Malades Hospital, Paris
  - Hôpitaux Universitaires de Strasbourg, Reference Center for Rare Disorders in Ophthalmic Genetics, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website, description of BrainPort Vision Pro — http://wicab.com